CLINICAL TRIAL: NCT04844008
Title: An Investigation of Whether Orally Delivered Nanobubbles Have a Physiological Effect on Joint Hypoxia?
Brief Title: Do Nanobubbles Improve Joint Hypoxia?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes in treatment pathway made recruitment unfeasible
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PID 15065
Record Dates: First submitted 2021-03-30; First posted 2021-04-14 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2021-03

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanobubble (Experimental): Sports drink nanobubble drink
  Interventions: Dietary Supplement: Nanobubble drink
- control (Placebo Comparator): Flavoured drink- no active ingredients
  Interventions: Dietary Supplement: Nanobubble drink

INTERVENTIONS:
Dietary Supplement: Nanobubble drink — Commercially available sports drink

SUMMARY:
Inflamed joints in patients with rheumatoid arthritis and psoriatic arthritis are characterized by low oxygen levels and inflammation. We propose to investigate whether tiny bubbles (nanobubbles) when given in a drink can alter oxygen level in joints. These nanobubbles are so small that they can enter the bloodstream when given as a drink. This information will give new information on the role of oxygen in joint inflammation and could possibly lead to new treatment approaches in the future.

ELIGIBILITY:
Inclusion Criteria:

* • Participant is willing and able to give informed consent for participation in the study.

  * Male or Female, aged 18 years or above.
  * Fulfil American College of Rheumatology/European League Against Rheumatism criteria (ACR/EULAR) 2010 Rheumatoid Arthritis Classification Criteria or fulfil Classification Criteria for Psoriatic Arthritis 2006 (CASPAR).
  * Selected joint for biopsy must be minimum Grade 2 synovial thickening for large joint (knee) and medium joint (wrist), or minimum Grade 3 synovial thickening for small joint (metacarpophalangeal).
  * Women of child bearing potential who are willing to use effective contraception (i.e. barrier, oral contraceptive pill, implanted contraception, or previous hysterectomy, bilateral oophorectomy) for the duration of the study.

Exclusion Criteria:

* • Currently on oxygen therapy.

  * Current enrolment in any other clinical study involving an investigational study treatment.
  * Pregnant or lactating, or women planning to become pregnant or initiating breastfeeding.
  * Intramuscular, intravenous or intra-articular administration of corticosteroid within 4 weeks prior to baseline visit.
  * Oral corticosteroid > 10 mg/day prednisolone or equivalent within 4 weeks prior to baseline visit.
  * Oral corticosteroid dose not stable for at least 4 weeks prior to baseline visit.
  * Oral non-steroidal anti-inflammatory drugs (including aspirin > 75 mg/ day and selective-cyclooxygenase inhibitors) dose not stable for at least 4 weeks prior to baseline visit.
  * Disease modifying anti-rheumatic drugs (DMARDs) dose not stable for at least 4 weeks prior to baseline visit.
  * History of septic arthritis.
  * Participants on warfarin, heparin, low molecular weight heparin, direct oral anticoagulants. Oral anti-platelet agents are permitted.
  * History of haemophilia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Change in Synovial fluid pO2 | Change in synovial fluid pO2 between day 1 and day 28

SECONDARY OUTCOMES:
Change in hypoxia-inducible factor 1α (HIF-1α) protein levels in synovial tissues | Change in hypoxia-inducible factor 1α (HIF-1α) protein between day 1 and day 28
Treatment Satisfaction Questionnaire for Medication (C) | Day28
  Validated PRO assessing: side effects, effectiveness, convenience and global satisfaction

OTHER OUTCOMES:
Change from baseline in the absolute and relative cell count in synovial fluid and synovial biopsy | day 28
Change from baseline of synovial fibroblast protein expression | day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No